CLINICAL TRIAL: NCT04909307
Title: Surveillance of Peripheral Blood Lymphocyte Subsets , Immune Function and Associations With Prognosis and Readiness of Return-to-work of CNS Germ Cell Tumor Survivors
Brief Title: Surveillance of Association of Immune Status and Prognosis of CNS Germ Cell Tumor Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chengcheng Guo (Other)
Responsible Party: Sponsor-Investigator, Chengcheng Guo, PhD, MD, Principal Investigator, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: ChengchengGuo
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Intracranial Germ Cell Tumor; Intracranial Germ Cell CNS Tumor, Childhood; Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: FDA-regulated Drug: No

SUMMARY:
Platinum-based chemotherapy, alternating at 21-days intervals with cycles of ifosfamide, cisplatin, and etoposide (ICE) and subsequently received radiotherapy were considered as standard treatment for intracranial germ cell tumors. However, whether reliable clinical data can quantify the damage degree of immunologic function caused by chemotherapy and radiotherapy is still unknown. This project regards the level of lymphocyte and immunocyte in peripheral blood as a quantitative index to reflect the dynamic change of the immunologic function of patients with CNS germ cell tumors before and after chemoradiotherapy treatment. Meanwhile, the investigators will also investigate the relationship between the level of lymphocyte and immunocyte in peripheral blood and the response rate of therapy.This study is designed to prospectively analyze the dynamic changes of immune status, prognosis and society function after standard treatment in patients with intracranial germ cell tumor.

DETAILED DESCRIPTION:
Immune status influences the reaction of anti-tumor and health condition of intracranial germ cell tumor patients. Peripheral blood and cerebrospinal fluid lymphocytes subsets, cytokines reflects those and be measured. Therefore, we designed the study to estimate patients health condition and survival outcomes in order to provides diversified assessment methods.

Peripheral blood will be collected from patients who will undergo surgery and/or neoadjuvant or adjuvant chemoradiotherapy. The setting time is before chemoradiotherapy, finishing chemoradiotherapy, pre-operation, postoperative day 1, day 3, day 5, and day 7. These blood samples will be used for detection and analysis in lymphocyte and immunocyte by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of an intracranial germ cell tumor (Histologically confirmed intracranial non-germinomatous or germinoma germ cell tumor).
* Histologically unconfirmed pineal and/or suprasellar tumors with serum/CSF beta HCG levels greater than 50 mIU/mL or AFP levels greater than 10 ng/ml or above institutional norm.
* No history of anti-tumor treatment
* Female subjects of childbearing potential have a negative pregnancy test and must agree to take effective contraceptive measures during the study period and within 3 months after the last dose;
* Be willing and able to provide written informed consent/assent for the trial

Exclusion Criteria:

* Patients with immune function deficiency : immunosuppression status, including autoimmune disease, post-operation of organ transplantation, in-taking immunosuppressive drug, human immunodeficiency virus (HIV) positive patients,
* Known history of active tuberculosis not adequately treated or positive QuantiFERON TB Gold test.
* Hypoproteinemia (eg, in case of severe liver disease or nephrotic syndrome) with serum albumin <3.0 g/dL.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with intracranial germ cell tumors and received anti-tumor therapy, including chemotherapy and radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between level of immune function and overall survival in patients with intracranial germ cell tumors. | 6 months
  Patients with intracranial germ cell tumors will be followed, prospectively from the time of discharge using review of the electronic medical record and as local guidance permits, phone calls at 3 and 6 months. The investigators will determine the associations between level of immune function after anti-tumor treatment and the objective remission rate and survival outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No